CLINICAL TRIAL: NCT04217174
Title: A Mobile Phone Intervention Using a Relational Human Talking Avatar to Promote Multiple Stages of the HIV Care Continuum in African American MSM
Brief Title: An Avatar-based Mobile Phone Intervention to Promote Health in African American MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Mississippi Medical Center (Other); Emory University (Other); Ruth M. Rothstein CORE Center (Other)
Responsible Party: Principal Investigator, Mark S Dworkin, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-1184; R01MH116721 (NIH)
Record Dates: First submitted 2019-12-31; First posted 2020-01-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Medication Adherence; Retention in Care
Keywords: HIV; adherence; retention in care; avatar; mobile phone application; food safety
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Avatar intervention app (Experimental): The intervention is a mobile phone app that features a realistic talking human avatar who promotes adherence to ART and retention in care, motivates, and provides information and opportunities for HIV care-related behavioral skills.
  Interventions: Behavioral: My Personal Health Guide
- Control app (Other): The control app is a mobile phone app that features a realistic talking human avatar who primarily promotes food safety and also offers knowledge of sugar content in food. This app is expected to have no effect on ART adherence and retention in care, however, it has never been tested to determine if it may have any effect so it has been categorized as Other (arm type) rather than as placebo.
  Interventions: Behavioral: My Personal Food Guide

INTERVENTIONS:
Behavioral: My Personal Health Guide — My Personal Health Guide is a theory-based mobile phone app that uses an Avatar as a personal health guide to increase patient knowledge of HIV disease and its complications and rationale for healthy behavior, increase self-efficacy and motivate participants to improve retention in care and medication adherence, and explain and illustrate behavioral skills related to retention in care, and adherence, with a result of improved behavior that leads to personal and population benefits through viral suppression and decreased risk of transmission, respectively. The relational aspect of the Avatar may be a powerful supplement to clinical care. The Avatar can encourage healthy behavior, acknowledge stigma and speak with empathy, audibly teach persons with low literacy, employ credible culturally appropriate phrasing, and invite the user to hear advice and motivational stories of other HIV-positive people and caregivers.
  Arms: Avatar intervention app
Behavioral: My Personal Food Guide — My Personal Food Guide is a mobile phone app that contains a talking realistic avatar who teaches about food safety, sugar content in selected foods, and some other food related information. The avatar motivates safe food behavior in order reduce the likelihood of food poisoning and promotes a healthy diet.
  Arms: Control app

SUMMARY:
The investigators propose to determine the efficacy of "My Personal Health Guide," a theory-based innovative talking relational human Avatar mobile phone application to engage HIV-positive AAMSM in adherence and retention in care. Providing an empathetic talking Avatar source of HIV-related information, motivation, and behavioral skills that is as private and convenient as their own mobile phone might produce a high impact by overcoming barriers to HIV adherence and retention in care such as stigma and health literacy.

DETAILED DESCRIPTION:
This proposal focuses on an innovative theory-driven intervention aimed at helping to improve outcomes for AAMSM targeting 3 stages of the HIV Care Continuum, (1) retention, (2) adherence to antiretroviral medication, and (3) viral suppression. My Personal Health Guide is an innovative talking relational human Avatar mobile phone application to engage HIV-positive AAMSM in adherence and retention in care. Development of this app was informed by the Information Motivation Behavioral Skills Model that focuses on feedback between information and motivation that affect one's behavioral skills, behaviors, and desired health outcomes. In the privacy of the user's home or anywhere they have their phone, the Avatar can encourage healthy behavior, acknowledge stigma and speak with empathy, audibly teach persons with low literacy, employ credible culturally appropriate phrasing, and invite the user to hear advice and motivational stories of other HIV-positive people and their caregivers. As part of a collaboration between UIC, Emory University, and the University of Mississippi Medical Center, the investigators propose to test the efficacy of the My Personal Health Guide Avatar application for young HIV-positive AAMSM. In this study, 250 HIV-positive AAMSM between the ages of 18-34 years with detectable viral load at baseline will be randomized to the My Personal Health Guide Avatar application or a food safety Avatar application control intervention for a 6-month period. Wirelessly monitored ART adherence will be collected for 1-month at baseline and then wirelessly monitored ART adherence, viral load, and clinic appointment data will be collected throughout the 6-month follow-up period. The investigators hypothesize that participants in the My Personal Health Guide intervention will demonstrate significant improvements in ART adherence, viral load, and retention in care during the follow-up period compared to control participants. The investigators will also identify mobile phone application functions that are associated with improvement in adherence in order to inform refinement of the application. The investigators hypothesize that more frequent use of Avatar information functions that included motivational messages will be associated with improved ART adherence.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported African American MSM
* 18 to 34 years old
* Smartphone owners
* Prescribed ART
* Have a viral load detectable within the past 4 weeks or self-reported or provider-reported history of adherence or treatment engagement problems.
* Participants may be initiating ART or already on ART.

Exclusion Criteria:

* Cannot speak English
* Decline to participate
* Participated in the usability and Beta testing phase of the app refinement that preceded this RCT
* Do not have a routine clinic appointment scheduled during the observation time.

Ages: 18 Years to 34 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a study of men who have sex with men so it is male gender based. Participants will self-report as male gender.
Enrollment: 315 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Viral suppression | From study enrollment until 2 months after study conclusion (9 months).
  The investigators will review medical records for HIV viral load measurements including the detectable measurement at study entry and all measurements that occur during the 6 months of follow-up and 2 months after. To ensure a high proportion of subjects have a follow-up viral load for comparison to their study entry viral load, the investigators will collect a fingerprick dried blood spot for viral load at the follow-up interview.

SECONDARY OUTCOMES:
Antiretroviral therapy adherence | 6 months before enrollment through two months after study conclusion (15 months).
  The investigators will use the Wisepill real-time electronic monitoring adherence device. The device obtains daily adherence information that can be analyzed as 7 monthly adherence measurements (1 month baseline and 6 months follow-up) calculated as proportion of doses taken out of days in the month. To supplement this measure, in the follow-up questionnaire the investigators will also collect the number of missed doses during the past month by self-report.
Retention in care | From app installation until study conclusion (6 months).
  To measure retention in care, the investigators will query participant's medical record to determine the number of HIV-related visits during the 6-months of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dworkin, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will depend on the nature of the request, available resources to fulfill the request, and IRB restrictions.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication in a peer-reviewed journal of the results of the three study aims, depending on the nature of the request, available resources to fulfill the request, and IRB restrictions, a dataset of deidentified data could be made available, estimated June 2025
Access Criteria: Request of PI with rationale.

REFERENCES:
- [Background] Dworkin MS, Lee S, Chakraborty A, Monahan C, Hightow-Weidman L, Garofalo R, Qato DM, Liu L, Jimenez A. Acceptability, Feasibility, and Preliminary Efficacy of a Theory-Based Relational Embodied Conversational Agent Mobile Phone Intervention to Promote HIV Medication Adherence in Young HIV-Positive African American MSM. AIDS Educ Prev. 2019 Feb;31(1):17-37. doi: 10.1521/aeap.2019.31.1.17. PMID 30742481
- [Background] Dworkin M, Chakraborty A, Lee S, Monahan C, Hightow-Weidman L, Garofalo R, Qato D, Jimenez A. A Realistic Talking Human Embodied Agent Mobile Phone Intervention to Promote HIV Medication Adherence and Retention in Care in Young HIV-Positive African American Men Who Have Sex With Men: Qualitative Study. JMIR Mhealth Uhealth. 2018 Jul 31;6(7):e10211. doi: 10.2196/10211. PMID 30064971
- [Result] Dworkin MS, Herrera K, Upton S, Luc CM, Jones J, Liu L, Jimenez A, Burns P, Ren R, Lee S, Woody M, Garofalo R. Evidence of Efficacy of the My Personal Health Guide Mobile Phone App on Antiretroviral Therapy Adherence Among Young African American Men Who Have Sex With Men at 1 Month: Randomized Controlled Trial. JMIR Mhealth Uhealth 2026;14:e75005. URL: https://mhealth.jmir.org/2026/1/e75005/ doi: 10.2196/75005
- [Derived] Dworkin MS, Herrera K, Upton S, Luc CM, Jones J, Burns P, Liu L, Jimenez A, Ren R, Woody M, Garofalo R, Lee S. Evidence of Efficacy of the My Personal Health Guide Mobile Phone App on Antiretroviral Therapy Adherence Among Young African American Men Who Have Sex With Men at 1 Month: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2026 Feb 3;14:e75005. doi: 10.2196/75005. PMID 41632958